CLINICAL TRIAL: NCT06261047
Title: Radiotherapy Delays Second-line Drug Therapy for Oligo Progressive Primary Liver Cancer: a Multicenter, Single-arm, Phase II Clinical Trial.
Brief Title: Radiotherapy Delays Second-line Drug Therapy for Oligo Progressive Primary Liver Cancer
Status: Recruiting | Type: Observational
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, jinbo Yue, Shandong Cancer Hospital and Institute
Other Study IDs: SDZLEC2023-389-02
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma; Radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: radiotherapy — radiotherapy

SUMMARY:
Recent years have seen significant advancements in the treatment landscape of advanced hepatocellular carcinoma (HCC), with the emergence of targeted and immunotherapy strategies reshaping first-line therapy. Sorafenib, a multi-targeted tyrosine kinase inhibitor, initially set the standard, followed by approvals for lenvatinib, regorafenib, cabozantinib, and ramucirumab. Immunotherapy, particularly combinations like atezolizumab with bevacizumab, has shown superior efficacy over sorafenib. Despite these advances, second-line therapies offer limited progression-free survival (mPFS: 2-3 months), necessitating new approaches. Radiotherapy, bolstered by technological advancements, has shown promise. Techniques like stereotactic body radiotherapy (SBRT) combined with PD-1 inhibitors achieve significant response rates and survival benefits. Combining radiotherapy with targeted immunotherapy has also demonstrated improved outcomes. Radiotherapy, especially in oligometastatic HCC, is increasingly favored due to its ability to enhance local control without increasing toxicity. These developments underscore the evolving landscape of HCC treatment towards personalized and multimodal approaches.

DETAILED DESCRIPTION:
hepatocellular carcinoma, stage IIIb, oligo progression

ELIGIBILITY:
Inclusion Criteria:

* Obtain written informed consent before implementing any trial-related procedures.
* Male or female, aged 18 years or older, and 75 years or younger.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1.
* Histological or cytological confirmation of primary hepatocellular carcinoma (HCC), or diagnosed according to the Clinical Diagnosis and Treatment Guidelines for Primary - Liver Cancer (2019 edition) issued by the National Health Commission of the People's Republic of China.
* Tumor staged as BCLC stage C; patients have ≤5 lesions (≤3 affected organs) with oligometastasis or oligoprogression.
* Liver function assessed by Child-Pugh score ≤7 points.
* Availability of tumor samples for biomarker assessment.
* Stable disease with systemic therapy for ≥3 months and an anticipated survival period of ≥6 months.

Exclusion Criteria:

* Diagnosis of malignancy other than liver cancer within 3 years before enrollment (excluding curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, and/or in situ carcinoma).
* Currently participating in interventional clinical research treatment, or received other investigational drugs or investigational device therapy within the past 4 weeks before enrollment.
* Received traditional Chinese medicine or immunomodulatory drugs with anti-tumor indications within 2 weeks before enrollment (including thymosin, interferon, interleukin, except for local use to control pleural effusion).
* Experienced active autoimmune diseases requiring systemic treatment (such as disease-modifying drugs, corticosteroids, or immunosuppressive agents) within 2 years before enrollment. Alternative therapies (such as thyroid hormone, insulin, or physiological glucocorticoids used for adrenal or pituitary insufficiency) are not considered systemic treatment.
* Received radiotherapy within 2 weeks before enrollment.
* HIV +
* Active untreated hepatitis B (defined as HBsAg positive with HBV-DNA copy number exceeding the upper limit of normal value in the laboratory of the participating center).
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma, stage IIIB, oligo progress
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 1 year
  The time from the initiation of radiotherapy until disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall response rate | 1 year
  the proportion of patients whose tumor size decreases (partial response) or disappears (complete response) following radiation
Overall survial | 1 year
  The time from the initiation of dignosis until death.
Disease control rate | 1 year
  the proportion of patients whose tumor size decreases (partial response) or disappears (complete response) or standard following radiation
Duration of control | 1 year
  the time of patients whose tumor size decreases (partial response) or disappears (complete response) or standard following radiation

CONTACTS AND LOCATIONS:
Overall Officials: jibo yue, dorctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Jinbo Yue, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hepatocellular carcinoma. Nat Rev Dis Primers. 2021 Jan 21;7(1):7. doi: 10.1038/s41572-021-00245-6. No abstract available. PMID 33479233
- [Result] Lee S, Kang TW, Song KD, Lee MW, Rhim H, Lim HK, Kim SY, Sinn DH, Kim JM, Kim K, Ha SY. Effect of Microvascular Invasion Risk on Early Recurrence of Hepatocellular Carcinoma After Surgery and Radiofrequency Ablation. Ann Surg. 2021 Mar 1;273(3):564-571. doi: 10.1097/SLA.0000000000003268. PMID 31058694
- [Result] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Result] Bruix J, Qin S, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Breder V, Gerolami R, Masi G, Ross PJ, Song T, Bronowicki JP, Ollivier-Hourmand I, Kudo M, Cheng AL, Llovet JM, Finn RS, LeBerre MA, Baumhauer A, Meinhardt G, Han G; RESORCE Investigators. Regorafenib for patients with hepatocellular carcinoma who progressed on sorafenib treatment (RESORCE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Jan 7;389(10064):56-66. doi: 10.1016/S0140-6736(16)32453-9. Epub 2016 Dec 6. PMID 27932229
- [Result] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Derived] Wang H, Zhang X, Zhu K, Jiang S, Liu T, Feng R, Dou X, Xu L, He J, Shi F, Yue J. Efficacy and safety of radiotherapy to delay second-line systemic therapy in patients with oligoprogressive hepatocellular carcinoma: study protocol of a multicentre, single-arm, phase II trial. Ther Adv Med Oncol. 2025 Apr 23;17:17588359251334538. doi: 10.1177/17588359251334538. eCollection 2025. PMID 40297623